CLINICAL TRIAL: NCT02361086
Title: A Phase 1/2 Open-Label, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Once-Daily VT-464 in Patients With Castration-Resistant Prostate Cancer
Brief Title: A Study to Evaluate Once-Daily Oral VT-464 in Patients With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innocrin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INO-VT-464-CL-004
Record Dates: First submitted 2015-01-29; First posted 2015-02-11 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Castration-resistant Prostate Cancer; CRPC
Keywords: castration-resistant prostate cancer; CYP17; P450c17a; lyase
MeSH Terms: interventions — VT-464

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Regimen 1: 7dayPM+DT (Experimental): VT-464: given orally once daily in 28 day cycles. Dosing in the evening before bed 7-days a week with a 2-week dose titration.
  Interventions: Drug: VT-464: given orally once daily in 28 day cycles
- Regimen 2: 7dayPM-DT (Experimental): VT-464: given orally once daily in 28 day cycles. Dosing in the evening before bed 7-days a week without dose titration.
  Interventions: Drug: VT-464: given orally once daily in 28 day cycles
- Regimen 3: 7dayAM+DT (Experimental): VT-464: given orally once daily in 28 day cycles. Dosing in the morning 7-days a week with a 2-week dose titration.
  Interventions: Drug: VT-464: given orally once daily in 28 day cycles
- Regimen 4: 7dayAM-DT (Experimental): VT-464: given orally once daily in 28 day cycles.Dosing in the morning 7-days a week without dose titration.
  Interventions: Drug: VT-464: given orally once daily in 28 day cycles
- Regimen 5: 5dayPM-DT (Experimental): VT-464: given orally once daily in 28 day cycles.Dosing in the evening before bed 5-days a week without dose titration.
  Interventions: Drug: VT-464: given orally once daily in 28 day cycles
- Regimen 6: 5dayAM-DT (Experimental): VT-464: given orally once daily in 28 day cycles.Dosing in the morning 5-days a week without dose titration.
  Interventions: Drug: VT-464: given orally once daily in 28 day cycles

INTERVENTIONS:
Drug: VT-464: given orally once daily in 28 day cycles — VT-464: given orally once daily in 28 day cycles either 5 days or 7 days a week.
  Other Names: VT-464

SUMMARY:
The goal of this clinical study is to determine the safety, tolerability, pharmacokinetics and activity of once-daily (QD) oral dosing of VT-464, a lyase-selective inhibitor of CYP17, in patients with castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a Phase 1/2 study of VT-464 in chemotherapy-naïve CRPC patients who are treatment-naive or who have failed prior therapy with abiraterone and/or enzalutamide. The study will examine several parallel QD dosing regimens of VT-464 using a traditional modified "3+3" Fibonacci study design. Approximately 3 dose-levels of VT-464 will be examined in each dosing regimen that is fully enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have documented histological or cytological evidence of adenocarcinoma of the prostate.
* Patients must have a minimum serum PSA level of >2 ng/ml that is rising based on the Prostate Cancer Working Group 2 criteria.
* Patients must have castrate levels of testosterone (<50 ng/dl [1.74 nmol/l]).
* Patients must have undergone orchiectomy, or have been on LHRH agonists or antagonists, for at least 3 months prior to study entry. Patients on LHRH agonists/antagonists must remain on these agents for the duration of the study.
* Patients must have an ECOG Performance Score of 0 or 1.

Key Exclusion Criteria:

* Patients who have received prior cytotoxic chemotherapy for castration-resistant prostate cancer unless enrolled in a previous chemotherapy cohort.
* Patients who have received second-line antihormonal therapy, including ketoconazole, aminoglutethimide, or high-dose estrogen within 30 days of study entry.
* Patients who have completed sipuleucel-T (Provenge ®) treatment within 30 days of study entry.
* Patients who have received TOK-001 (Galeterone®) or any other investigational product directed towards the androgen receptor or androgen biosynthesis.
* Patients who have received antiandrogens such as flutamide (EULEXIN®), bicalutamide (CASODEX®), or nilutamide (NILANDRON®) for > 3 months must be off treatment for 6 weeks and demonstrate a continued rise in PSA after withdrawal. Patients on antiandrogens for < 3 months must be off medication for 2 weeks. Patients on 5 alpha reductase inhibitors such as finasteride (PROSCAR®, PROPECIA®), or dutasteride (AVODART®) must stop medication at least 3 months from study entry.
* Patients who require pharmacological or replacement doses of systemic corticosteroids or who have received systemic corticosteroids within 30 days of study entry; use of topical, inhaled or ophthalmic steroids is permitted.
* Patients who have received palliative radiotherapy within 4 weeks of study entry.
* Patients with a history within the last 3 years of another invasive malignancy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of VT-464 by evaluating adverse events, vital signs, physical examination findings, concomitant medications and laboratory tests. | The first 28-day continuous dosing cycle at target dose.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of VT-464 | After the first dose of VT-464
Area under the plasma concentration versus time curve (AUC) of VT-464 | After the first dose of VT-464
Time to maximum plasma concentration (Tmax) of VT-464 | After the first dose of VT-464

OTHER OUTCOMES:
The change in PSA from baseline using waterfall plots in response to VT-464 | At least monthly over the first 8 28-day dosing cycles
Objective tumor response to VT-464 at the end of even-numbered cycles using RECIST 1.1 criteria | At least every other month over the first 8 28-day dosing cycles
The absolute and percent change from baseline in adrenal, pituitary, and testicular hormone concentrations in response to VT-464 | At least monthly over the first 8 28-day dosing cycles

CONTACTS AND LOCATIONS:
Overall Officials: Joel Eisner, Study Director — Innocrin Pharmaceutical
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Urology Cancer Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Virginia Oncology Associates, Norfolk, Virginia